CLINICAL TRIAL: NCT02081079
Title: A Phase 2, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination in Treatment-Naive and Treatment-Experienced Subjects With Chronic Genotype 4 or 5 HCV Infection
Brief Title: Efficacy and Safety of Ledipasvir/Sofosbuvir Fixed-Dose Combination in Treatment-Naive and Treatment-Experienced Subjects With Chronic Genotype 4 or 5 HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1119; 2013-003978-27 (EudraCT Number)
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2016-04

CONDITIONS: Chronic Genotype 4 HCV; Chronic Genotype 5 HCV
Keywords: HCV GT 4; HCV GT 5
MeSH Terms: interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Genotype 4 (Experimental): LDV/SOF for up to 12 weeks in treatment-naive and treatment-experienced participants with genotype 4 hepatitis C virus (HCV) infection
  Interventions: Drug: LDV/SOF
- Genotype 5 (Experimental): LDV/SOF for up to 12 weeks in treatment-naive and treatment-experienced participants with genotype 5 hepatitis C virus (HCV) infection
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — LDV/SOF (90/400 mg) FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
This study is to evaluate the efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) in participants with chronic genotype 4 or 5 hepatitis C virus (HCV) infection as measured by the proportion of subjects with sustained virologic response (SVR12), defined as HCV RNA < lower limit of quantification (LLOQ) 12 weeks after discontinuation of therapy.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA ≥ 10^4 IU/mL at screening
* Chronic genotype 4 or 5 HCV Infection
* Individuals may be treatment naive or treatment experienced
* Presence or absence of cirrhosis, a liver biopsy may be required
* Healthy according to medical history and physical examination with the exception of HCV diagnosis
* Agree to use two forms of highly effective contraception for the duration of the study

Exclusion Criteria:

* History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the individual's participation for the full duration of the study or not be in the best interest of the individual in the opinion of the investigator
* Prior exposure to approved or experimental HCV specific direct acting antiviral(s) (DAA) other than NS3/4A protease inhibitors
* History of any other clinically significant chronic liver disease
* Evidence of or history of decompensated liver disease
* HIV or chronic hepatitis B (HBV) infection
* Hepatocellular carcinoma (HCC) or other malignancy (with exception of certain resolved skin cancers)
* Chronic use of immunosuppressive agents or immunomodulatory agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Kersey, MSc, Study Director — Gilead Sciences
Locations (5):
- France (5):
  - Clermont-Ferrand
  - Clichy
  - Limoges
  - Toulouse
  - Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Abergel A, Metivier S, Samuel D, Jiang D, Kersey K, Pang PS, Svarovskaia E, Knox SJ, Loustaud-Ratti V, Asselah T. Ledipasvir plus sofosbuvir for 12 weeks in patients with hepatitis C genotype 4 infection. Hepatology. 2016 Oct;64(4):1049-56. doi: 10.1002/hep.28706. Epub 2016 Jul 29. PMID 27351341
- [Derived] Abergel A, Asselah T, Metivier S, Kersey K, Jiang D, Mo H, Pang PS, Samuel D, Loustaud-Ratti V. Ledipasvir-sofosbuvir in patients with hepatitis C virus genotype 5 infection: an open-label, multicentre, single-arm, phase 2 study. Lancet Infect Dis. 2016 Apr;16(4):459-64. doi: 10.1016/S1473-3099(15)00529-0. Epub 2016 Jan 21. PMID 26803446

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in France. The first participant was screened on 07 March 2014. The last study visit occurred on 17 February 2015.
Pre-assignment Details: 91 participants were screened.
Groups:
- Genotype 4: Ledipasvir/sofosbuvir (Harvoni®; LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet administered orally once daily for up to 12 weeks in participants with genotype 4 hepatitis C virus (HCV) infection
- Genotype 5: LDV/SOF (90/400 mg) FDC tablet administered orally once daily for up to 12 weeks in participants with genotype 5 HCV infection
Period: Overall Study
Arm/Group | Genotype 4 | Genotype 5
Started | 44 | 41
Completed | 40 | 39
Not Completed | 4 | 2
Not completed — Lack of Efficacy | 3 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were enrolled and received at least 1 dose of study drug
Groups:
- Genotype 4: Treatment-naive: LDV/SOF (90/400 mg) FDC tablet administered orally once daily for up to 12 weeks in treatment-naive participants with genotype 4 HCV infection
- Genotype 4: Treatment-experienced: LDV/SOF (90/400 mg) FDC tablet administered orally once daily for up to 12 weeks in treatment-experienced participants with genotype 4 HCV infection
- Genotype 5: Treatment-naive: LDV/SOF (90/400 mg) FDC tablet administered orally once daily for up to 12 weeks in treatment-naive participants with genotype 5 HCV infection
- Genotype 5: Treatment-experienced: LDV/SOF (90/400 mg) FDC tablet administered orally once daily for up to 12 weeks in treatment-experienced participants with genotype 5 HCV infection
- Total: Total of all reporting groups
Arm/Group | Genotype 4: Treatment-naive | Genotype 4: Treatment-experienced | Genotype 5: Treatment-naive | Genotype 5: Treatment-experienced | Total
Number analyzed (Participants) | 22 | 22 | 21 | 20 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (9.2) | 50 (8.8) | 61 (10.4) | 64 (8.6) | 57 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 10 | 10 | 36
  Male | 11 | 17 | 11 | 10 | 49
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3 | 5 | 0 | 0 | 8
  White | 19 | 17 | 21 | 20 | 77
Region of Enrollment [Number; unit: participants]
  France | 22 | 22 | 21 | 20 | 85
HCV RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 6.0 (0.40) | 6.3 (0.48) | 6.2 (0.48) | 6.6 (0.39) | 6.3 (0.48)
HCV Genotype [Number; unit: participants]
  Genotype 4 | 22 | 22 | 0 | 0 | 44
  Genotype 5 | 0 | 0 | 21 | 20 | 41
Cirrhosis Status [Number; unit: participants]
  Absence | 21 | 13 | 18 | 14 | 66
  Presence | 1 | 9 | 3 | 6 | 19
IL28b Status [Number; unit: participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 7 | 1 | 13 | 6 | 27
    CT | 11 | 16 | 7 | 11 | 45
    TT | 4 | 5 | 1 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants with genotype 4 or 5 HCV infection who were enrolled and received at least on dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 4: Treatment-naive | Genotype 4: Treatment-experienced | Genotype 5: Treatment-naive | Genotype 5: Treatment-experienced
Number analyzed (Participants) | 22 | 22 | 21 | 20
percentage of participants | 95.5 | 90.9 | 95.2 | 95.0

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued LDV/SOF Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: participants were enrolled and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- Genotype 4: LDV/SOF (90/400 mg) FDC tablet administered orally once daily for up to 12 weeks in participants with genotype 4 HCV infection
Arm/Group | Genotype 4 | Genotype 5
Number analyzed (Participants) | 44 | 41
percentage of participants | 0 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 4: Treatment-naive | Genotype 4: Treatment-experienced | Genotype 5: Treatment-naive | Genotype 5: Treatment-experienced
Number analyzed (Participants) | 22 | 22 | 21 | 20
percentage of participants
  SVR4 | 95.5 | 90.9 | 95.2 | 95.0
  SVR24 | 95.5 | 90.9 | 95.2 | 95.0

4. Secondary Outcome: Percentage of Patients With Virologic Failure
Description: Virologic failure was defined as either:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment); or
  * Relapse:
    * HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while receiving treatment
Time Frame: Up to posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 4: Treatment-naive | Genotype 4: Treatment-experienced | Genotype 5: Treatment-naive | Genotype 5: Treatment-experienced
Number analyzed (Participants) | 22 | 22 | 21 | 20
percentage of participants
  On-treatment Virologic Failure | 0 | 0 | 0 | 0
  Relapse | 4.5 | 9.1 | 4.8 | 5.0

5. Secondary Outcome: Change From Baseline in HCV RNA at Weeks 2, 4, 8, and 12
Time Frame: Baseline; Weeks 2, 4, 8, and 12
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Genotype 4: Treatment-naive | Genotype 4: Treatment-experienced | Genotype 5: Treatment-naive | Genotype 5: Treatment-experienced
Number analyzed (Participants) | 22 | 22 | 21 | 20
log10 IU/mL
  Change at Week 2 | -4.65 (0.397) | -4.77 (0.495) | -4.97 (0.479) | -4.94 (0.477)
  Change at Week 4 | -4.86 (0.396) | -5.17 (0.490) | -5.07 (0.474) | -5.39 (0.381)
  Change at Week 8 | -4.88 (0.401) | -5.18 (0.484) | -5.07 (0.474) | -5.45 (0.387)
  Change at Week 12 | -4.88 (0.401) | -5.18 (0.484) | -5.07 (0.474) | -5.45 (0.387)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set: participants were randomized and received at least 1 dose of study drug
Arm/Group | Genotype 4 | Genotype 5
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/41
Other Adverse Events (participants affected / at risk) | 31/44 | 31/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotype 4 (N=44) | Genotype 5 (N=41)
Depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Genotype 4 (N=44) | Genotype 5 (N=41)
Vertigo (Ear and labyrinth disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 4 | 1
Asthenia (General disorders) | 10 | 16
Fatigue (General disorders) | 9 | 4
Nasopharyngitis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 3
Wound (Injury, poisoning and procedural complications) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 11 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years